CLINICAL TRIAL: NCT07320274
Title: ArcFlex Sheath in TAVR Trial(Arc-FIT)
Brief Title: ArcFlex Sheath in TAVR Trial
Acronym: Arc-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Arc-FIT trial
Record Dates: First submitted 2025-09-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Valve Disease, Aortic
Keywords: TAVR; Sheath; ArcFlex
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ArcFlex Sheath (Experimental): ArcFlex Sheath
  Interventions: Device: ArcFlex Sheath
- control group (Placebo Comparator): The ordinary sheath
  Interventions: Device: ordinary sheath

INTERVENTIONS:
Device: ArcFlex Sheath — TAVR is a crucial treatment method for aortic valve diseases. The requirements for the device to cross the aortic arch and for the bioprosthetic valve to be coaxial are quite high, and they are key steps for the success of the surgery. Investigators' aim is to evaluate the safety and effectiveness of a variable-bend sheath for the TAVR procedure.
  Arms: ArcFlex Sheath
Device: ordinary sheath — ordinary sheath
  Arms: control group

SUMMARY:
TAVR is a crucial treatment method for aortic valve diseases. The requirements for the device to cross the aortic arch and for the bioprosthetic valve to be coaxial are quite high, and they are key steps for the success of the surgery. Investigators' aim is to evaluate the safety and effectiveness of a variable-bend sheath for the TAVR procedure.

ELIGIBILITY:
Inclusion Criteria:

* Judged by a professional cardiologist to require TAVR surgery
* NYHA ≥ II grade
* Evaluated by the cardiac team, the peripheral vascular approach is suitable for performing the surgery via the femoral route
* Expected lifespan is greater than 1 year (5) Patients who can understand the purpose of the trial, voluntarily participate, sign the informed consent form, and are willing to undergo relevant examinations and clinical follow-ups.

Exclusion Criteria:

* Presence of other valvular diseases requiring concurrent intervention.
* Anatomical characteristics unsuitable for transcatheter valve implantation.
* Severe mitral stenosis due to organic causes requiring surgical valve replacement or repair.
* Hypertrophic obstructive cardiomyopathy (unexplained myocardial hypertrophy >1.5 cm).
* Acute myocardial infarction within the past 30 days.
* Intracardiac mass, thrombus, or vegetation indicated by echocardiography.
* Active infective endocarditis or any other active infection.
* Intolerance to tolerate anticoagulant or antiplatelet therapy.
* Coagulopathy or refusal to receive blood transfusion therapy.
* Known allergy to device materials or contrast agents.
* Acute peptic ulcer or gastrointestinal bleeding within the past 3 months.
* Stroke or transient ischemic attack (TIA) within the past 3 months.
* Requirement for emergency surgical treatment for any reason.
* Expected life expectancy of less than 12 months due to non-cardiac causes.
* Severe disabling dementia or inability to perform activities of daily living.
* Participation in other clinical trials of drugs or medical devices prior to enrollment and not yet reached the primary endpoint of that study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
surgical instruments | 24 hours
  The success rate of immediate surgical instruments

SECONDARY OUTCOMES:
30-day mortality rate | 30days
  30-day mortality rate
One-year mortality rate | 1 year
  One-year mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mao Y, Liu Y, Zhai M, Jin P, Chen F, Yang Y, Zhu G, Yang T, Zhang G, Xu K, Shang X, Zhao Y, Ni B, Li H, Tang M, Jian Z, Yang Y, Zhang H, Wei L, Liu J, Noterdaeme T, Lange R, Guo Y, Pan X, Wu Y, Yang J. Clinical value of aortic arch morphology in transfemoral TAVR: artificial intelligence evaluation. Int J Surg. 2025 Mar 1;111(3):2338-2347. doi: 10.1097/JS9.0000000000002232. PMID 39869394